CLINICAL TRIAL: NCT03746418
Title: Effect of Addition of Dexmedetomidine During Ultrasound Guided Bilateral Single Shot Erector Spinae Plane Block in Patients Undergoing Posterior Lumbar Interbody Fusion Under General Anesthesia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: mona bologh elmorad,MD (Unknown); mohmed naser shaddad,MD (Unknown)
Responsible Party: Principal Investigator, Ahmed Said Elgebaly,MD, director, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: tantaESB
Record Dates: First submitted 2018-11-11; First posted 2018-11-19 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Double Level Lumbar Spondylolisthesis (L3-L5); Posterior Lumbar Interbody Fusion (PLIF); Lumbar Fixation Surgery
Keywords: erector spinae; dexmedetomidine; ultrasound; lumbar interbody fusion; spondylolisthesis
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Placebo Comparator): received 20 ml of 0. 25% bupivacaine plus one mL normal saline bilaterally.
  Interventions: Drug: Ultrasound Guided Bilateral single shot Erector Spinae Plane Block
- Group II (Active Comparator): received 20 ml of 0.25% bupivacaine with supplementation of 1 mL containing 100µg dexmedetomidine bilaterally
  Interventions: Drug: Ultrasound Guided Bilateral single shot Erector Spinae Plane Block

INTERVENTIONS:
Drug: Ultrasound Guided Bilateral single shot Erector Spinae Plane Block — Under aseptic technique and after skin infiltration with 3 ml of 2% lidocaine, a 22G, 50-mm, insulated facet type needle (visioplex® - vygon - France) was introduced in plane in a cephalad to caudad direction until (L3) transverse process was hit [figure1(A)(B)(C)] and the needle was slightly withdrawn. The confirmation of the correct position of the needle tip was done by injecting 0.5-1 ml of LA. Once confirmed, 20 ml of the drug was administered under vision after confirming negative aspiration of blood. LA distribution was observed in both cranial and caudal directions. This was repeated on the other side also. Twenty minutes later, sensory loss to cold was evident between (T10-T 12) and (L5-S1) vertebral level of the posterior dermatomes and dermatomes of the anterior roots of the spinal nerves (lumbar plexus, upper leg) on both sides without hemodynamic changes. Motor function of the legs was evaluated with a Bromage (0-3) score.

SUMMARY:
Posterior lumbar interbody fusion (PLIF) is the management of choice in double level lumbar (L) spondylolisthesis (L3-L5) after ineffective conservative treatment. We evaluated bilateral ultrasound (US)-guided single shot erector spinae plane (ESP) block at the level of lumbar 3 (L3) vertebra with or without dexmedetomidine (Dex).

DETAILED DESCRIPTION:
Objectives: Posterior lumbar interbody fusion (PLIF) is the management of choice in double level lumbar (L) spondylolisthesis (L3-L5) after ineffective conservative treatment. We evaluated bilateral ultrasound (US)-guided single shot erector spinae plane (ESP) block at the level of lumbar 3 (L3) vertebra with or without dexmedetomidine (Dex).

Methods: A prospective controlled randomized, double-blind study comparing two groups of patients; each group included 20 patients of double level spondylolisthesis (L3-L5) scheduled for (PLIF) under general anesthesia combined with bilateral US-guided ESP single shot block at (L3). Group I received 20 ml of 0. 25% bupivacaine plus one mL normal saline bilaterally. Group II received 20 ml of 0.25% bupivacaine with supplementation of 1 mL containing 100µg dexmedetomidine bilaterally. Post-Anesthesia Care Unit (PACU) length of stay, the total dose of postoperative analgesics need, postoperative visual analogue score (VAS) at 1h, 6h, 12h, and 24 h after the operation and postoperative complications which related to block or opioids were recorded.

ESP block at combined with (Dex) is a safe, effective block with no complications. Addition of 100µg Dex to preoperative ESP block provided good postoperative opioid-sparing analgesia, facilitated the early emergence and shortened the length of stay in the PACU during (PLIF) for double level spondylolisthesis (L3-L5).

ELIGIBILITY:
Inclusion Criteria:

* belonged to the American Society of Anesthesiologists (ASA) physical status I or II
* either sex
* aged 18-60 years
* body mass index less 35 kg/m2
* complaining from double level lumbar spondylolisthesis (L3-L5)
* scheduled for elective surgical intervention aimed at lumbar spine fixation by PLIF - under general anesthesia.

Exclusion Criteria:

* obesity (body mass index > 35 kg/m2)
* infection of the skin at the site of the needle puncture
* allergies to either of the study drugs
* bleeding disorder
* and recent use of opioid.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
changes in Post-Anesthesia Care Unit (PACU) length of stay | at 1hours, 6hours, 12hours, and 24 hours after the operation
  assessment of changes in the Post-Anesthesia Care Unit (PACU) length of stay in (minutes) during the first 24 hours was reported.
changes in the total dose of postoperative analgesics need | at 1hours, 6hours, 12hours, and 24 hours after the operation
  assessment of changes in the total dose of postoperative analgesics need in the first 24 hours were reported.
changes in postoperative visual analogue score (VAS) | at 1hours, 6hours, 12hours, and 24 hours after the operation
  assessment of changes in the postoperative visual analogue score (VAS)in the first 24 hours was reported.
  Scoring and Interpretation: Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
  Based on the distribution of pain VAS scores in post-surgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm) . Normative values are not available. The scale has to be shown to the patient otherwise it is an auditory scale, not a visual one.
changes in recovery time | at 1hours, 6hours, 12hours, and 24 hours after the operation
  assessment of changes in the recovery time length in (minutes) during the first 24 hours was reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Said Elgebaly, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chaudhary NK, Singh S. Continuous ultrasound-guidederector spinae plane block for post-operative pain management in lumbar spine surgery: A case series. Indian J Anaesth. 2018 Aug;62(8):638-639. doi: 10.4103/ija.IJA_160_18. No abstract available. PMID 30166664
- [Result] Melvin JP, Schrot RJ, Chu GM, Chin KJ. Low thoracic erector spinae plane block for perioperative analgesia in lumbosacral spine surgery: a case series. Can J Anaesth. 2018 Sep;65(9):1057-1065. doi: 10.1007/s12630-018-1145-8. Epub 2018 Apr 27. PMID 29704223
- [Result] Zhang S, Ye C, Lai Q, Yu X, Liu X, Nie T, Zhan H, Dai M, Zhang B. Double-level lumbar spondylolysis and spondylolisthesis: A retrospective study. J Orthop Surg Res. 2018 Mar 16;13(1):55. doi: 10.1186/s13018-018-0723-3. PMID 29548343
- [Result] Adhikary SD, Bernard S, Lopez H, Chin KJ. Erector Spinae Plane Block Versus Retrolaminar Block: A Magnetic Resonance Imaging and Anatomical Study. Reg Anesth Pain Med. 2018 Oct;43(7):756-762. doi: 10.1097/AAP.0000000000000798. PMID 29794943